CLINICAL TRIAL: NCT02823847
Title: Non-invasive Oral Cancer Screening Among Individuals Who Have HIV Infection
Brief Title: Non Invasive Oral Cancer Screening Among HIV Infected Individuals
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Baylor College of Medicine (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2015-1030; NCI-2016-01073 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Malignant Neoplasms of Mesothelial and Soft Tissue; Human Immunodeficiency Virus
Keywords: Malignant neoplasms of mesothelial and soft tissue; Human immunodeficiency virus; HIV; Carbon monoxide test; Self-help materials; Visual Oral Screening Examination; Direct Fluorescent Oral Visualization Examination; Oral Biopsy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Screening (Experimental): Participants given a screening interview at baseline. Carbon monoxide testing given to participants at baseline. Participants who want to stop smoking are given referral information for a tobacco cessation program. Participants undergo an oral examination using conventional light, and oral examination using a fluorescence light-based hand held device at baseline, and again two weeks later. Oral lesions still present after two weeks are biopsied. Participants with premalignant and malignant oral lesions [PMOL]) given printed materials and web-based programs for tobacco and alcohol cessation.
  Interventions: Behavioral: Screening Interview; Device: Carbon Monoxide Test; Behavioral: Self-Help Materials; Procedure: Visual Oral Screening Examination; Procedure: Direct Fluorescent Oral Visualization Examination; Procedure: Oral Biopsy

INTERVENTIONS:
Behavioral: Screening Interview — Participants asked about demographic information, and questions about history of tobacco, alcohol, and mouthwash use. Interview lasts about 7 minutes.
Device: Carbon Monoxide Test — Carbon monoxide testing given to participants at baseline. Participants blow into a device that measures the amount of carbon monoxide in the lungs.
Behavioral: Self-Help Materials — Participants who want to stop smoking are given referral information for a tobacco cessation program at baseline.
  Participants with premalignant and malignant oral lesions [PMOL]) given printed materials and web-based programs for tobacco and alcohol cessation.
Procedure: Visual Oral Screening Examination — Intraoral exam performed under incandescent (white light) conditions at baseline, and again two weeks later.
Procedure: Direct Fluorescent Oral Visualization Examination — Intraoral exam performed under reduced room lighting with a handheld autofluorescence imaging device at baseline, and again two weeks later.
Procedure: Oral Biopsy — Premalignant and malignant oral lesions [PMOL]) still present 2 weeks after oral exam are biopsied.

SUMMARY:
The goal of this clinical research study is to learn how a new method for performing oral (mouth) exams can help doctors check for suspicious lesions (called premalignant and malignant oral lesions [PMOL]) in the mouth of HIV-infected smokers.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be asked to come to the clinic for 2 study visits.

First Study Visit:

* You will be asked questions about your history of tobacco, alcohol, and mouthwash use. You will also be asked questions about your demographic information (such as age, sex at birth, sexual orientation and gender identification, educational level, and insurance status). This interview will last about 7 minutes.
* You will be asked to blow into a device that measures the amount of carbon monoxide in your lungs. Smokers may have a larger amount of carbon monoxide in their lungs.
* You will be given referral information for a tobacco cessation program if you want help to stop smoking.

After this first interview, you will have a standard dental exam of your mouth and throat using normal office lighting. Any suspected PMOLs will be photographed. Right after that, a second dental exam will be performed, using a hand-held fluorescent light device. This device will be shined into your mouth to help the doctor check for PMOLs. Any suspected PMOLs will be photographed under the fluorescent light.

Second Study Visit (Follow-up):

About 2 weeks after your first study visit, you will be asked to return to the clinic. During this visit, you will have another oral exam with both standard and fluorescent light. You will also be asked 3 questions about being enrolled in any tobacco cessation programs. If any PMOL(s) that were found during the first visit are is still present, the study staff will collect a biopsy of the PMOL tissue. The type of biopsy you have will depend on the number of PMOLs you have and their location, size, shape, and appearance. To perform this biopsy, the affected area is removed by cutting it out (possibly completely). Local anesthesia will be used. The biopsied tissue samples will be sent to the laboratory for routine testing. The results of the biopsies will be used to test the accuracy of the 2 oral exams.

A dental appointment will be made with you about 7-14 days after the oral biopsy to inspect the wound and discuss the biopsy result.

Length of Study:

Your active study participation will be over after the second study visit.

This is an investigational study. The standard oral exams are performed using FDA-approved and commercially available methods. The use of the fluorescent light is considered investigational.

The performance of the PMOL follow-up biopsy is considered standard of care.

Up to 80 participants will be enrolled in this research study. All will be enrolled at Bering Omega Community Services Dental Clinic.

ELIGIBILITY:
Inclusion Criteria:

1. HIV positive individuals seeking dental care at Bering Omega/Houston Area Community Services
2. Being able to speak English and/or Spanish

Exclusion Criteria:

1. patients under 18 years of age
2. patients current participation in a tobacco cessation program
3. Patients unwilling or unable to provide consent
4. Patients declining oral biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Positive Predictive Value for Premalignant and Malignant oral lesions (PMOL) | 2 weeks
  Positive predictive value defined as the number of true positives (confirmed PMOLs) divided by the total number of suspicious lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Irene M. Tami-Maury, DRPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Bering Omega/Houston Area Community Services, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org